CLINICAL TRIAL: NCT01087437
Title: Testing the Effect of Crustacean's Gastrolith Nutraceutical on Mineralization Rate During Distraction Osteogenesis
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Collaborators: Amorfical (Unknown)
Responsible Party: Ron Lamdan, Hadassah Medical Organization
Allocation: Non-Randomized | Model: Single Group | Purpose: Treatment
Other Study IDs: LAM002-HMO-CTIL
Record Dates: First submitted 2010-03-14; First posted 2010-03-16 (Estimated); Last update posted 2014-04-01 (Estimated); Status verified 2014-03

CONDITIONS: Skeletal Deformities; Leg Length Discrepancy
Keywords: Distraction osteogenesis
MeSH Terms: conditions — Leg Length Inequality

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- gastrolith calcium treatment (Experimental)
  Interventions: Dietary Supplement: gastrolith calcium

INTERVENTIONS:
Dietary Supplement: gastrolith calcium

SUMMARY:
BACKGROUND: Distraction osteogenesis, the gradual lengthening of bones, is performed in order to equalize leg length discrepancy and correct skeletal deformities or to achieve greater height in short stature people. The femur and tibia are the bones most frequently lengthened. The surgery is currently performed at Hadassah Medical Center routinely by the pediatric orthopedic team utilizing a variety of external fixation devices.

The procedure involves application of an external fixation device to the bone, creation of an osteotomy and gradual, controlled distraction of the bone fragments On the last week of the distraction phase and every month thereafter, patients will be provided with a monthly supply of gastrolith calcium in a sealed container (65 capsules of 500 mg each, provided by Amorphical). Starting on the first day of the last week of the distraction phase, during the entire consolidation phase until the external fixator is removed; adults will orally consume two (2) 500 mg capsules a day (total of 1 gr of gastrolith calcium). Children will be given 25 mg calcium per kg body weight up to the daily adult dose of 1000mg .

ELIGIBILITY:
Inclusion Criteria:

1. Males and females
2. Ages 4-30 years old.

Exclusion Criteria:

1. Product Allergy
2. Refusal to participate the study.
3. Metabolic Disorders

Ages: 4 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 2011-01

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organizaton, Jerusalem, Israel